CLINICAL TRIAL: NCT00696137
Title: Open-label, Long-term Extension Study for Treatment of Breakthrough Cancer Pain With BEMA™ Fentanyl
Brief Title: Long-term Extension Study of BEMA™ Fentanyl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEN-290
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Depression
Keywords: Chronic Pain; Ventilatory Response to Hypercapnia (VRH)
MeSH Terms: conditions — Respiratory Insufficiency; Chronic Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEMA Fentanyl (Experimental): BEMA Fentanyl
  Interventions: Drug: BEMA Fentanyl

INTERVENTIONS:
Drug: BEMA Fentanyl — buccal soluble film; 200, 400, 600, 800, and 1200 mcg fentanyl; up to 4 times daily
  Other Names: bioerodible mucoadhesive; fentanyl buccal soluble film; ONSOLIS

SUMMARY:
This study is designed to provide continued access to BEMA Fentanyl for those subjects who previously participated in FEN-202 and who wish to continue using BEMA Fentanyl for the treatment of their breakthrough cancer pain.

DETAILED DESCRIPTION:
This was an open label, long-term, extension study designed to provide continued access to EMA Fentanyl to those patients with breakthrough cancer pain who were treated for at least 2 weeks in FEN-202, the long term safety study used for worldwide registration. Patients were followed in an outpatient setting. Use of BEMA Fentanyl and occurrence of serious adverse events (SAEs) were monitored. Throughout the study, all patients continued their background opioid regimen and were permitted to use their rescue medication if adequate pain relief was not realized within 30 minutes following application of BEMA Fentanyl.

ELIGIBILITY:
Inclusion Criteria:

1. previously qualified for and participated in study FEN-202 for at least 2 weeks,
2. wish to continue using BEMA Fentanyl for treatment of breakthrough pain episodes, and
3. provide signed informed consent at screening prior to any study procedures.

Exclusion Criteria:

1. they have developed a new medical condition after initial enrollment in FEN-202 which, in the opinion of the investigator, would preclude safe and appropriate use of BEMA Fentanyl or participation in this study, or
2. there is evidence of improper use of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, MD, Study Chair — BioDelivery Sciences International

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BEMA Fentanyl
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | BEMA Fentanyl
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Was Not Measured in This Study. The Number of Deaths in the Long Term Follow-up Will be Reported.
Description: Efficacy was not measured in this study as the intention was to evaluate long term safety in this population. The number of deaths in the long term follow-up will be reported.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BEMA Fentanyl
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events were not recorded in this study because non-serious AEs have already been assessed in FEN-201 and FEN-202.
Arm/Group | BEMA Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days